CLINICAL TRIAL: NCT06582394
Title: Effect of Virtual BASRD Reality Training Versus Conservative Treatment In Chronic Hemipretic Stroke Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/738
Record Dates: First submitted 2024-08-21; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exp Group (Experimental)
  Interventions: Combination Product: Exp Group
- Control Group (Active Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Combination Product: Exp Group — Balance and coordination were targeted through virtual stepping tasks, where participants practiced stepping in various directions to improve postural control and lower limb function. Additionally, they performed virtual balance exercises by standing on simulated platforms of varying stability. For gait and mobility, participants practiced walking in a virtual environment with real-time feedback to correct gait abnormalities. They also encountered virtual obstacles, which required them to adapt their walking patterns and improve mobility. In this study, both the intervention and control groups underwent a 6-week treatment plan consisting of 5 sessions per week, with each session lasting 45 minutes.
  Arms: Exp Group
Other: Control group — For gait training, participants practiced walking on flat surfaces, sometimes with the assistance of parallel bars or walking aids, to improve their walking speed, step length, and rhythm. They also performed sit-to-stand exercises to strengthen the lower limbs and improve mobility for daily activities. Additionally, manual therapy techniques, such as joint mobilizations and stretching, were applied to reduce spasticity and increase range of motion in the affected limbs. Both treatment groups progressed based on individual capabilities, with therapists adjusting exercises accordingly throughout the study. In this study, both the intervention and control groups underwent a 6-week treatment plan consisting of 5 sessions per week, with each session lasting 45 minutes.
  Arms: Control Group

SUMMARY:
In hemiparetic stroke patient's VR is very useful. Due to hemiparesis one side muscle weakness occurs because of disruption in brain, spinal cord and nervous system technologies improvs motor activities of patients, by improvement in motor activities patients perform activities in better way.

DETAILED DESCRIPTION:
The study's main aim is to check virtual reality's effect on conservative treatment in hemiparetic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Both ischemia and hemorrhagic stroke.
* Stroke Patients who were in Chronic phase diagnosed by Physician were included in the study.

Exclusion Criteria:

* Patient with the history of previous stroke attacks.
* Brainstem stroke
* Epilepsy
* Severely impaired communication and cognition
* Parkinson's disease and multiple sclerosis
* Other musculoskeletal and psychological disorder

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Barthel index | 12 Months
  The Barthel Index is a scale used to measure a person's ability to perform basic activities of daily living (ADL) independently. It assesses 10 areas of functioning, with a focus on mobility and self-care. Scores range from 0 to 100, with higher scores indicating greater independence. Stroke-Specific Quality of Life Scale (SS-QOL) It assesses the impact of stroke on the quality of life across various domains, including physical, emotional, social, and cognitive aspects. It uses 12 domains with items scored on a 5-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Depalpur, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No